CLINICAL TRIAL: NCT07289893
Title: Investigation of the Effects of Kettlebell Training on Pain, Function and Performance in Rotator Cuff-Related Shoulder Pain; Randomized Controlled Trial.
Brief Title: Investigation of the Effects of Kettlebell Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Turgut, Prof, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30.01.2024
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Pain; Rotator Cuff Injuries
Keywords: Kettlebell Exercises
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Kettlebell Exercise Group
  Interventions: Other: Kettlebell Exercise
- Control Group (Active Comparator): Standard Rehabilitation Group
  Interventions: Other: Standard Exercise

INTERVENTIONS:
Other: Kettlebell Exercise — 8-week Kettlebell Exercises compare with 8-week Standard Rehabilitation Program
  Arms: Exercise Group
Other: Standard Exercise — 8-week Standard Rehabilitation Program compare with 8-week Kettlebell Exercises
  Arms: Control Group

SUMMARY:
Kettlebell exercises are seen as one of the approaches that can be used conservatively in individuals with shoulder pain. However, it is still unknown what results it has on its therapeutic effects. These findings highlight the need for higher quality studies evaluating the effects of kettlebell use and exercises for shoulder pain. Therefore, the purpose of this study was to investigate the effects of 8 weeks of kettlebell training on shoulder pain, function, and performance.

The hypotheses of our study are as follows:

* H1: In individuals with Rotator Cuff-Related Shoulder Pain, the improvement in shoulder-related pain perception is greater with Kettlebell training compared to the standard rehabilitation program.
* H2: In individuals with Rotator Cuff Related Shoulder Pain, shoulder function improvement is greater with Kettlebell training compared to the standard rehabilitation program.
* H3: In individuals with Rotator Cuff-Related Shoulder Pain, shoulder performance improvement is greater with Kettlebell training than with the standard rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are willing to participate and have been doing licensed/unlicensed amateur or professional sports for at least 3 years,
* Individuals with Tegner Activity Scale ≥ 5,
* A history of shoulder pain of at least 6 weeks,
* At least 3 points measured using the 0 to 10 point Numerical Pain Scale (NPS),
* Shoulder pain that worsens with resisted shoulder flexion, abduction or external rotation,
* Rotator cuff tendinopathies,
* Tears smaller than 1 cm,
* Secondary shoulder instability without major trauma (due to rotator cuff muscle weakness, etc.)

Exclusion Criteria:

* History of fracture and/or surgery in the shoulder area,
* Adhesive capsulitis,
* Those with passive joint range of motion deficit,
* Individuals with a positive Apprehension Test and/or Sulcus Sign test and multidirectional shoulder instability,
* Numbness or tingling in the upper extremity with cervical compression test or upper extremity compression test,
* Systemic or neurological disease,
* Corticosteroid injection within 3 months before the intervention,
* Physical therapy in the 6 months before the intervention,
* Those with a history of dislocation and subluxation,
* Those who are pregnant,
* Those who did not participate in the study for 2 consecutive sessions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 0th and 8th Week
  It is a self-report questionnaire that measures pain and disability in the shoulder. It consists of 13 items in 2 subscales: pain (5 items) and disability (8 items). Items for both subscales are measured with visual analog scales ranging from 0 (no pain or difficulty) to 10 (worst pain imaginable or difficult enough to require assistance).
Seated Single-Arm Shot-Put Test | 0th and 8th Week
  Participants are placed in a position that does not restrict arm movement on the test side. In this position, they are instructed to hold a 3 kg ball in their hands at shoulder level with pain. Thus, from this initial positioning the participant pushes the ball as far as possible without noticing any compensation with the body. The evaluator administers the test independently and requests 3 applications at the participant's maximum capacity, with verbal stimulation and 1 minute rest between repetitions, and the average of these 3 applications is calculated.
Upper Extremity Y Balance Test | 0th and 8th Week
  For testing; The mechanism is established by combining 1.5 meter (m) lines in the medial, inferolateral and superolateral directions at appropriate angles. For the test, participants are asked to come into a push-up position and reach in all three directions with their free hands. Maximum reach distance will be recorded in centimeters (cm). In order to normalize the reach distances according to the limb length, the maximum values in each direction are summed, divided by 3 times the limb length and multiplied by 100.
Closed Kinetic Chain Upper Extremity Stability Test | 0th and 8th Week
  Individuals will be positioned in a push-up position with their bodies aligned in a straight line when viewed from the side, with a distance of 90 cm between their hands. Athletes will be asked to touch the dominant hand to the dorsum of the other hand within 15 seconds, and the total number of repetitions is recorded. The tests are repeated three times with a 45-second rest between tests and the average of the results is recorded.
Evaluation of Shoulder Isometric Muscle Strength | 0th and 8th Week
  Values resulting from isometric contraction will be recorded in kg. Muscle strength measurements will be evaluated bilaterally, in three repetitions, for 5 seconds. The average value of the triplicate results obtained will be recorded.
Evaluation of Hand Grip Strength | 0th and 8th Week
  Measurements were made while the individuals were standing, with the elbow and wrist in full extension. Measurements are repeated three times at 5-second intervals on the dominant and non-dominant hands (first right, then left and right again, etc.) and recorded in kilograms, and then their average is taken.

SECONDARY OUTCOMES:
Global Rating of Change (GROC) | 0th and 8th Week
  This scale is a frequently used scale for the evaluation of clinical research in the musculoskeletal field. It is used to determine the improvement or deterioration of patients over a specified period of time. On the numerical scale, one represents "my pain has decreased a lot in a good way," while seven means "my pain has increased a lot in a bad way," and people report changes in pain compared to baseline.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University, Ankara
  - Fenerbahce University, Istanbul

IPD SHARING:
Plan to Share IPD: No